CLINICAL TRIAL: NCT02378623
Title: PARADOX Trial: A Prospective, Double-Blind, Randomized Controlled Trial in Patients With Patent Foramen Ovale and Endocardial Device Leads on Apixaban for Prevention of Paradoxical Emboli
Brief Title: Patients With Patent Foramen Ovale and Endocardial Device Leads on Apixaban for Prevention of Paradoxical Emboli
Acronym: PARADOX
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew funding - May 2016
Sponsor: Mayo Clinic (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Christopher V. DeSimone, M.D., Ph.D., PI, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-008633
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Patent Foramen Ovale; Cardiac Implantable Electronic Device
Keywords: paradoxical embolism; lead thrombus; ICD; Pacemaker; Cognitive decline; Stroke; TIA
MeSH Terms: conditions — Foramen Ovale, Patent; Embolism, Paradoxical; Cognitive Dysfunction; Stroke | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Active Comparator): Intervention group: Apixaban 5 mg by mouth two times daily in addition to usual medical therapy (or 2.5 mg two times daily for subjects who fulfilled any 2 of the following criteria: age≥80 years, body weight≤60kg, and/or serum creatinine≥1.5 mg/dL). Planned treatment duration is 2 years
  Interventions: Drug: Apixaban
- Placebo (Placebo Comparator): Control group: Matched placebo by mouth two times daily in addition to usual medical therapy. Planned treatment duration is 2 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban — Patients who meet the study eligibility criteria and consent for enrollment will be randomized in a 1:1 ratio to intervention with apixaban or control group with placebo. The randomization will be performed by a computer generated block randomization protocol. Randomization will be stratified according to pre-existing CIED (≥6 months) vs. new implantation (<6 months from date of implant), in order to ensure at least 25% of patients have longstanding lead placement.
  Other Names: Eliquis
  Arms: Apixaban
Drug: Placebo — Patients who meet the study eligibility criteria and consent for enrollment will be randomized in a 1:1 ratio to intervention with apixaban or control group with placebo. The randomization will be performed by a computer generated block randomization protocol. Randomization will be stratified according to pre-existing CIED (≥6 months) vs. new implantation (<6 months from date of implant), in order to ensure at least 25% of patients have longstanding lead placement.
  Arms: Placebo

SUMMARY:
Patients with a patent foramen ovale in the setting of endocardially placed cardiac implantable electronic devices such as pacemakers, defibrillators, or resynchronization therapies are likely at higher risk for paradoxical embolic events from device lead thrombus. The investigators are conducting this study to determine if the anticoagulant medication Apixaban is more effective at reducing MRI detected brain lesions compared to placebo.

DETAILED DESCRIPTION:
This is a prospective, double-blinded, placebo-controlled, randomized controlled trial (RCT).

400 patients who meet the study eligibility criteria and consent for enrollment will be randomized in a 1:1 ratio to intervention with apixaban or control group with placebo. The randomization will be performed by a computer generated block randomization protocol. The majority of patients will begin intervention with Apixaban or placebo at the time of cardiac device placement (n approximately 300), and at least a quarter of the randomized patients (n ≥100) will include preexisting CIED (≥6 months) in place. Each patient will undergo a baseline MRI and a comprehensive cognitive screening examination. Repeat MRI and cognitive assessment will be performed at a follow-up period of two years from date of randomization (or less if clinical stroke/TIA occurs prior to this follow-up period). All subjects will receive a phone call at 6 months, 12 months, and 18 months post-randomization to assess for endpoints and adverse events, as well as changes in clinical status, medications, and to assess study medication compliance.

ELIGIBILITY:
Inclusion:

* A clinical indication for a trans venous pacemaker, ICD, or CRT device, or presence of a pre-existing endovascular CIED
* Presence of a PFO (regardless of shunt direction) confirmed with trans-esophageal or trans-thoracic echocardiography with color flow Doppler and/or agitated saline
* Absence of any contraindication for anticoagulation
* Absence of a clinical indication for systemic anticoagulation
* Ability to give informed consent for the trial
* Able to undergo head MRI and consent for MRI study to be performed in presence of CIED

Exclusion:

* Patients with a survival expectancy of less than one year
* Patients who require systemic anticoagulation for any established clinical indication (excluding the presence of PFO with CIED)
* Patients with an atrial or ventricular septal defect that is hemodynamically significant and requires repair as suggested by the ACC/AHA 2008 guidelines on evaluation and treatment of adult congenital heart diseases
* Absence of a CIED or no clinical indication for a trans venous CIED
* Contraindication to undergoing an MRI
* Patients with an active infection that cannot be treated successfully prior to randomization
* Women who are pregnant or breastfeeding, or women of child-bearing potential who do not wish to use an effective method of birth control during the course of study in a manner such that the risk of failure is minimized
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s)
* Known sensitivity to any of the active substances or their excipients to be administered during dosing with study medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Increase in number of new brain lesions detected on MRI ≥3 mm in size at 2 years post-baseline MRI (or earlier if premature termination of study follow-up). | 2 years
  The primary objective of this study is to determine whether medical therapy with apixaban lowers the rate of new MRI cerebral lesions compared to placebo in pacemaker, defibrillator, and resynchronization device therapy recipients with a PFO

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Asirvatham, MD, Principal Investigator — Mayo Clinic; Christopher DeSimone, MD, Principal Investigator — Mayo Clinic; Paul Friedman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States